CLINICAL TRIAL: NCT00666211
Title: Phase III Randomized Trial of an Opioid Titration Order Sheet Compared to Standard of Care in Patients With Cancer Related Pain.
Brief Title: Opioid Titration Order Sheet or Standard Care in Treating Patients With Cancer Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Nancy Wells, Research Professor of Nursing; Director, VUMC Nursing; Researcher, Vanderbilt-Ingram Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: VICC SUPP 0424; P30CA068485 (NIH); VU-VICC-SUPP-0424; VU-VICC-040410
Record Dates: First submitted 2008-04-23; First posted 2008-04-24 (Estimated); Results first posted 2012-09-06 (Estimated); Last update posted 2012-09-06 (Estimated); Status verified 2012-08

CONDITIONS: Brain and Central Nervous System Tumors; Chronic Myeloproliferative Disorders; Leukemia; Lymphoma; Lymphoproliferative Disorder; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Neoplasms; Pain; Precancerous Condition; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: pain; unspecified adult solid tumor, protocol specific; accelerated phase chronic myelogenous leukemia; acute undifferentiated leukemia; adult acute lymphoblastic leukemia in remission; adult acute myeloid leukemia in remission; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); atypical chronic myeloid leukemia, BCR-ABL negative; blastic phase chronic myelogenous leukemia; chronic myelomonocytic leukemia; chronic phase chronic myelogenous leukemia; mast cell leukemia; meningeal chronic myelogenous leukemia; progressive hairy cell leukemia, initial treatment; prolymphocytic leukemia; recurrent adult acute lymphoblastic leukemia; recurrent adult acute myeloid leukemia; recurrent adult T-cell leukemia/lymphoma; refractory chronic lymphocytic leukemia; refractory hairy cell leukemia; relapsing chronic myelogenous leukemia; secondary acute myeloid leukemia; stage I adult T-cell leukemia/lymphoma; stage I chronic lymphocytic leukemia; stage II adult T-cell leukemia/lymphoma; stage II chronic lymphocytic leukemia; stage III adult T-cell leukemia/lymphoma; stage III chronic lymphocytic leukemia; stage IV adult T-cell leukemia/lymphoma; stage IV chronic lymphocytic leukemia; T-cell large granular lymphocyte leukemia; stage I adult Hodgkin lymphoma; stage II adult Hodgkin lymphoma; stage III adult Hodgkin lymphoma; stage IV adult Hodgkin lymphoma; anaplastic large cell lymphoma; angioimmunoblastic T-cell lymphoma; cutaneous B-cell non-Hodgkin lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; stage I cutaneous T-cell non-Hodgkin lymphoma; stage II cutaneous T-cell non-Hodgkin lymphoma; stage III cutaneous T-cell non-Hodgkin lymphoma; stage IV cutaneous T-cell non-Hodgkin lymphoma; recurrent mycosis fungoides/Sezary syndrome; stage I mycosis fungoides/Sezary syndrome; stage II mycosis fungoides/Sezary syndrome; stage III mycosis fungoides/Sezary syndrome; stage IV mycosis fungoides/Sezary syndrome; adult grade III lymphomatoid granulomatosis; adult nasal type extranodal NK/T-cell lymphoma; Waldenstrom macroglobulinemia; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma; contiguous stage II adult Burkitt lymphoma; contiguous stage II adult diffuse large cell lymphoma; contiguous stage II adult diffuse mixed cell lymphoma; contiguous stage II adult diffuse small cleaved cell lymphoma; contiguous stage II adult immunoblastic large cell lymphoma; contiguous stage II adult lymphoblastic lymphoma; contiguous stage II grade 1 follicular lymphoma; contiguous stage II grade 2 follicular lymphoma; contiguous stage II grade 3 follicular lymphoma; contiguous stage II mantle cell lymphoma; contiguous stage II marginal zone lymphoma; stage I adult Burkitt lymphoma; stage I adult diffuse large cell lymphoma; stage I adult diffuse mixed cell lymphoma; stage I adult diffuse small cleaved cell lymphoma; stage I adult immunoblastic large cell lymphoma; stage I adult lymphoblastic lymphoma; stage I grade 1 follicular lymphoma; stage I grade 2 follicular lymphoma; stage I grade 3 follicular lymphoma; stage I mantle cell lymphoma; stage I marginal zone lymphoma; stage I small lymphocytic lymphoma; noncontiguous stage II adult Burkitt lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult diffuse small cleaved cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult lymphoblastic lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; noncontiguous stage II mantle cell lymphoma; noncontiguous stage II marginal zone lymphoma; noncontiguous stage II small lymphocytic lymphoma; stage III adult Burkitt lymphoma; stage III adult diffuse large cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III mantle cell lymphoma; stage III marginal zone lymphoma; stage III small lymphocytic lymphoma; stage IV adult Burkitt lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV mantle cell lymphoma; stage IV marginal zone lymphoma; stage IV small lymphocytic lymphoma; recurrent adult Burkitt lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult grade III lymphomatoid granulomatosis; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; intraocular lymphoma; primary central nervous system non-Hodgkin lymphoma; primary central nervous system Hodgkin lymphoma; post-transplant lymphoproliferative disorder; chronic eosinophilic leukemia; chronic neutrophilic leukemia; primary myelofibrosis; essential thrombocythemia; polycythemia vera; extramedullary plasmacytoma; isolated plasmacytoma of bone; monoclonal gammopathy of undetermined significance; stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma; primary systemic amyloidosis; refractory multiple myeloma; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; myelodysplastic/myeloproliferative neoplasm, unclassifiable; recurrent adult Hodgkin lymphoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Myeloproliferative Disorders; Leukemia; Lymphoma; Lymphoproliferative Disorders; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Pain; Precancerous Conditions; Leukemia, Myeloid, Accelerated Phase; Leukemia, Biphenotypic, Acute; Congenital Abnormalities; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Blast Crisis; Leukemia, Myelomonocytic, Chronic; Leukemia, Myeloid, Chronic-Phase; Leukemia, Mast-Cell; Leukemia, Prolymphocytic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Hairy Cell; Leukemia, Large Granular Lymphocytic; Hodgkin Disease; Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Lymphoma, T-Cell, Cutaneous; Mycosis Fungoides; Sezary Syndrome; Lymphoma, Extranodal NK-T-Cell; Waldenstrom Macroglobulinemia; Lymphoma, B-Cell, Marginal Zone; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Intraocular Lymphoma; Pdgfra-Associated Chronic Eosinophilic Leukemia; Leukemia, Neutrophilic, Chronic; Primary Myelofibrosis; Thrombocythemia, Essential; Polycythemia Vera; Monoclonal Gammopathy of Undetermined Significance; Immunoglobulin Light-chain Amyloidosis | interventions — Early Intervention, Educational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard of Care (Active Comparator): Standard pain control drugs.
  Interventions: Other: educational intervention; Other: questionnaire administration
- Opioid Titration (Experimental): Pain will be Monitored and Medication Titrated
  Interventions: Other: educational intervention; Other: Titrated pain management; Other: questionnaire administration

INTERVENTIONS:
Other: educational intervention — Participants will be educated on pain management.
Other: Titrated pain management — Pain will be Monitored and Medication Titrated
  Arms: Opioid Titration
Other: questionnaire administration — Participants will be given questionnaires to complete.

SUMMARY:
RATIONALE: An Opioid Titration Order Sheet that allows healthcare providers to adjust the dose and schedule of pain medication may help improve pain treatment for patients with cancer. It is not yet known whether the use of an Opioid Titration Order Sheet is more effective than standard care in treating pain caused by cancer.

PURPOSE: This randomized phase III trial is studying an Opioid Titration Order Sheet to see how well it works compared with standard care in treating patients with cancer pain.

DETAILED DESCRIPTION:
OBJECTIVES:

* To examine the effect of an opioid titration order sheet on pain outcomes.
* To examine the effect of an opioid titration order sheet on secondary outcomes of function, mood, and quality of life.

OUTLINE: This is a multicenter study. Participating centers are randomized to 1 of 2 treatment arms.

* Arm I (usual care): After completion of baseline assessments, patients undergo a standardized pain education program over approximately 15 minutes. The program consists of standard written materials about communicating pain to providers, opioids and side effect management, as well as a tailored discussion about patient concerns and specific information about prescribed opioid medications. Patients are also instructed in the use of the daily pain diary. Patients are then discharged from the clinic with instructions to contact the treating physician (through standard procedures) for problems with pain or side effects. The study staff conducts weekly telephone interviews to prevent changes in patient pain management practice. The treating physician continues to manage pain in their usual manner.
* Arm II (opioid titration order sheet): After completion of baseline assessments, patients undergo the standardized pain education program and are instructed in the use of the daily pain diary as described in arm I. The treating physician signs an Opioid Titration Order Sheet (OTOS) providing a baseline dose and schedule. The OTOS is faxed to study staff and verified. Patients are then discharged from the clinic with instructions to contact the research nurse for problems with pain or side effects. The treating physician also contacts the study staff if he/she is made aware of any problems pertaining to the patient's pain control. The research nurse, in consultation with study physician, manages pain according to the OTOS and manages opioid side effects using standing orders. Referral to the treating physician is made as needed.

Patients' pain is managed on study for 8 weeks in the absence of unacceptable toxicity, pain crisis, or new site of pain.

Patients complete a demographic questionnaire at baseline and other questionnaires at 2, 4, and 6 weeks (over the telephone) and at 8 weeks (at site or by telephone), including the Functional Assessment Screening Questionnaire (FASQ), the Brief Pain Inventory-Interference (PPI-I), The Profile of Mood States-Short Form (POMS-SF), and the Quality of life (FACT-G) questionnaire. Patients also complete a pain diary recording daily measures of pain dimensions, analgesic use (i.e., fixed dose opioids, rescue doses, and non-opioids), adjuvant medications, and side effects that prevented the patient from taking medications. Data in the pain diary is transcribed over the telephone on a weekly basis.

Clinical data, including the type of cancer, stage of disease, time since diagnosis, current treatment for cancer, type of pain, time since onset of pain, and time of first opioid prescription, as well as information regarding analgesics (opioid and non-opioid), adjuvant medications, and medications to manage side effects prescribed during the study is collected from patients' medical records. Anticancer and palliative treatment received during the study is monitored via treating physician records.

The physician charts are reviewed after study completion to determine whether pain, treatment, and response are adequately documented and treated. The documentation in the physician charts is compared to the documentation obtained by the study staff during the study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed carcinoma
* Cancer-related pain requiring fixed-dose opioid therapy

  * Has received ≥ 1 week of fixed-dose opioid therapy AND meets any of the following criteria:

    * Inadequate pain control as defined by the patient
    * Requires 2 or more rescue doses per day
    * Requires adjustments in pain regimen (either fixed or breakthrough dosing)
* No pain crisis that requires hospitalization or immediate anesthetic or neurosurgical intervention
* No predominantly neuropathic pain (e.g., peripheral neuropathy) as assessed by the treating physician

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* ANC > 1,500/mm³
* Platelet count > 100,000/mm³
* Serum bilirubin < 1.5 mg/dL
* Serum creatinine < 2.5 mg/dL
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Nutritional, pulmonary, and cardiac status must be considered adequate to tolerate the proposed study therapy
* Must be available for active follow-up
* No documented active psychiatric disorder (i.e., psychosis or major depression) that would preclude informed consent or the patient's ability to comply with study procedures
* No significant infection
* No concerns about compliance with medication regimens or medical follow-up
* No excessive alcohol use

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Concurrent chemotherapy or radiotherapy allowed

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2005-05; Primary Completion 2010-01 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Wells, DNSc, RN, Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (11):
- United States (11):
  - Jennie Stuart Medical Center, Hopkinsville, Kentucky
  - Mitchell Memorial Cancer Center at Owensboro Medical Health System, Owensboro, Kentucky
  - Erlanger Health System, Chattanooga, Tennessee
  - Tennessee Plateau Oncology, Crossville, Tennessee
  - Center for Biomedical Research, Knoxville, Tennessee
  - The Jones Clinic, Memphis, Tennessee
  - Vanderbilt-Ingram Cancer Center - Cool Springs, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center at Franklin, Nashville, Tennessee
  - Meharry Medical College, Nashville, Tennessee
  - Veterans Affairs Medical Center - Nashville, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study opened to accrual May 2005 through May 2010. Although 99 patients were consented one was determined ineligible, thus only 98 went on study.
Period: Overall Study
Arm/Group | Standard of Care | Opioid Titration
Started | 42 | 56
Completed | 22 | 18
Not Completed | 20 | 38
Not completed — Withdrawal by Subject | 10 | 13
Not completed — went off medication, no more pain | 1 | 0
Not completed — patient non-compliant | 6 | 6
Not completed — disease progression | 1 | 8
Not completed — Lost to Follow-up | 2 | 0
Not completed — toxicity | 0 | 2
Not completed — hospital admission | 0 | 5
Not completed — Death | 0 | 2
Not completed — off tx for other complicating disease | 0 | 1
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care | Opioid Titration | Total
Number analyzed (Participants) | 42 | 56 | 98
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 33 | 49 | 82
  >=65 years | 9 | 7 | 16
Age Continuous [Mean (Standard Deviation); unit: years] | 55.6 (1) | 56.4 (1) | 56 (1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 20 | 39
  Male | 23 | 36 | 59
Region of Enrollment [Number; unit: participants]
  United States | 42 | 56 | 98

OUTCOME MEASURES:

1. Primary Outcome: Pain Intensity
Description: Patients in each arm will each have 9 measures: daily scores averaged over 1 week with baseline to week 8:
  1. Average daily pain intensity 0 (no pain) to 10 (worst) scale
  2. Worst daily pain intensity 0 (no pain) to 10 (worst) scale
Time Frame: Baseline(Week 0) to week 8, Total time frame is 9 weeks.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard of Care | Opioid Titration
Number analyzed (Participants) | 42 | 56
units on a scale
  Average Daily Pain Intensity | 5.60 (2.76) | 6.44 (1.89)
  Worst Daily Pain Intensity | 5.11 (2.45) | 5.98 (1.96)

2. Secondary Outcome: Ability to Engage in Activities of Daily Living (ADL)
Description: The Functional Assessment Screening Questionnaire (FASQ) scale is used, scored at baseline and at weeks 2, 4, 6, 8. The FASQ consists of 15 questions about ability to perform ADL with minimum score of 1 (easy to perform) to a maximum score of 5 (N/A, meaning someone else performs this activity for the patient or else the patient chooses not to do it). A summary mean score is generated with a minimum score of 1 and a maximum score of 5.
Time Frame: Baseline(Week 0) to week 8, Total time frame is 9 weeks.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard of Care | Opioid Titration
Number analyzed (Participants) | 42 | 56
units on a scale
  Baseline | 2.18 (0.61) | 1.99 (0.58)
  Week 2 | 2.14 (0.73) | 2.06 (0.67)
  Week 4 | 1.94 (0.57) | 1.91 (0.55)
  Week 6 | 2.01 (0.73) | 2.03 (0.49)
  Week 8 | 1.98 (0.67) | 1.96 (0.58)

3. Secondary Outcome: Interference in Daily Life Due to Pain
Description: Patients in each arm will each have 5 measures on the Brief Pain Inventory (BPI) scale: baseline + weeks 2, 4, 6, 8. The BPI consists of 7 questions about interference of pain in daily life, answered on a scale of 0 (does not interfere) to 10 (completely interferes). The summary score is the average from the 7 questions, with higher score indicating greater interference due to pain.
Time Frame: 9 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard of Care | Opioid Titration
Number analyzed (Participants) | 42 | 56
units on a scale
  Baseline | 4.49 (2.54) | 4.23 (2.30)
  Week 2 | 4.25 (2.89) | 4.12 (2.26)
  Week 4 | 4.16 (2.82) | 3.48 (2.03)
  Week 6 | 3.78 (2.99) | 3.16 (2.21)
  Week 8 | 3.01 (2.43) | 3.68 (2.42)

4. Secondary Outcome: Mood Disturbance
Description: Patients in each arm will each have 5 measures on the Profile of Mood States-Short Form (POMS-SF): baseline + weeks 2, 4, 6, 8. The POMS-SF consists of 37 questions, querying 6 mood states (anxiety, depression, anger, confusion, fatigue, and vigor), with responses on a scale from 0 (not at all) to 4 (extremely). To generate a summary score, questions on vigor state are first recoded to reverse the scale, so that higher summary scores consistently indicate greater mood disturbance.
Time Frame: 9 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard of Care | Opioid Titration
Number analyzed (Participants) | 42 | 56
units on a scale
  Baseline | 1.48 (0.55) | 1.21 (0.63)
  Week 2 | 1.45 (0.63) | 1.20 (0.52)
  Week 4 | 1.37 (0.70) | 1.12 (0.52)
  Week 6 | 1.19 (0.64) | 1.22 (0.66)
  Week 8 | 1.14 (0.58) | 1.32 (0.70)

5. Secondary Outcome: Quality of Life
Description: Each patient in each arm is scored on the Functional Assessment of Cancer Therapy-General (FACT-G) at baseline + week 8 with 4 related sub-scales (physical, social/family, emotional, functional well-being. To generate sub-scale scores, physical and emotional items are reverse coded & items are then summed, such that higher values indicate better quality of life. Thus, each sub-scale score ranges from 0 (not at all, worse outcome) to 4 (very much, better outcome) with a minimum total score of 0 (worst quality of life) to a maximum of 16 (good quality of life).
Time Frame: 9 weeks
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Standard of Care | Opioid Titration
Number analyzed (Participants) | 42 | 56
scores on a scale
  Physical at baseline | 1.94 (0.83) | 2.11 (0.77)
  Physical at week 8 | 2.18 (0.93) | 2.34 (0.86)
  Social/family at baseline | 3.02 (0.82) | 3.30 (0.77)
  Social/family at week 8 | 3.03 (0.90) | 2.88 (0.92)
  Emotional at baseline | 2.55 (0.90) | 2.93 (0.69)
  Emotional at week 8 | 2.88 (0.77) | 2.42 (0.83)
  Functional well-being at baseline | 1.81 (0.92) | 1.75 (0.82)
  Functional well-being at week 8 | 1.88 (0.86) | 1.88 (0.78)

6. Primary Outcome: Pain-related Distress
Description: Patients in each arm will each have 9 measures: daily scores averaged over 1 week with baseline to week 8. Pain-related distress scale is from 0 (no pain) to 10 (worst pain).
Time Frame: Baseline(Week 0) to week 8, Total time frame is 9 weeks.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard of Care | Opioid Titration
Number analyzed (Participants) | 42 | 56
units on a scale | 3.32 (2.50) | 4.87 (2.64)

7. Primary Outcome: Pain Duration
Description: Pain duration in hours 0 to 24
Time Frame: at 9 weeks
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Standard of Care | Opioid Titration
Number analyzed (Participants) | 42 | 56
hours | 8.40 (6.06) | 11.31 (7.78)

ADVERSE EVENTS:
Arm/Group | Standard of Care | Opioid Titration
Serious Adverse Events (participants affected / at risk) | 1/42 | 8/56
Other Adverse Events (participants affected / at risk) | 13/42 | 27/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard of Care (N=42) | Opioid Titration (N=56)
Somnolence/depressed level of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Pain - Throat/pharynx/larynx - odynophagia (General disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Death not associated with CTCAE term (General disorders) | 0 (0) | 1 (1)
nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
infection with normal ANC (Infections and infestations) | 0 (0) | 1 (1)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pain - Back (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
extremity-lower gait (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Mucositis/stomatisis (Gastrointestinal disorders) | 0 (0) | 2 (2)
aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
neutrapenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
hyponatremia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
weight loss (Investigations) | 0 (0) | 1 (1)
dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
fatigue (General disorders) | 0 (0) | 1 (1)
confusion (Psychiatric disorders) | 0 (0) | 1 (1)
Ventricular arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Infection with unknown ANC (Infections and infestations) | 0 (0) | 1 (1)
fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard of Care (N=42) | Opioid Titration (N=56)
drowsiness, somnolence (Nervous system disorders) | 4 (13) | 2 (9)
confusion (Psychiatric disorders) | 2 (4) | 1 (12)
anorexia (Psychiatric disorders) | 2 (15) | 0 (0)
bruising (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
cardiac arrhythmia (Cardiac disorders) | 2 (2) | 1 (3)
constipation (Gastrointestinal disorders) | 1 (8) | 4 (41)
cough (Respiratory, thoracic and mediastinal disorders) | 2 (5) | 2 (13)
dysphagia (Nervous system disorders) | 0 (0) | 4 (33)
edema (General disorders) | 0 (0) | 4 (14)
fatigue (General disorders) | 0 (0) | 8 (46)
nausea (Gastrointestinal disorders) | 0 (0) | 6 (50)
neuropathy (Nervous system disorders) | 1 (2) | 3 (11)
pain, extremity (Musculoskeletal and connective tissue disorders) | 3 (10) | 0 (0)
dysgeusia (Nervous system disorders) | 2 (7) | 0 (0)
Dysarthria (Nervous system disorders) | 3 (18) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes